CLINICAL TRIAL: NCT04060030
Title: Treatment of Social and Language Deficits With Leucovorin for Young Children With Autism
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: Autism Speaks (Other); State University of New York - Downstate Medical Center (Other)
Responsible Party: Principal Investigator, Richard Frye, Principal Investigator, Southwest Autism Research & Resource Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AS Leucovorin
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Language Disorders
MeSH Terms: conditions — Autism Spectrum Disorder; Language Disorders | interventions — Leucovorin

STUDY DESIGN:
Intervention Model Description: Prospective randomized 12-week double-blind placebo-controlled study followed by 12-week open label
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple masking during blinded phase, followed by unblinding during open label phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-leucovorin calcium (Experimental): The liquid form of leucovorin calcium will be dosed by weight, with a target dose of 1mg/kg/day, divided into two daily doses. This product may be taken alone or mixed with liquid. Participants randomized to this arm will receive active treatment for both 12-week phases of the study.
  Interventions: Drug: Levoleucovorin Calcium
- Placebo (Placebo Comparator): The placebo will mimic the experimental treatment in flavor, odor, packaging, and dosing instructions. Participants randomized to this arm will receive placebo for the first 12 weeks of the study, then active treatment for the remaining 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levoleucovorin Calcium — Liquid leucovorin calcium dosed by weight
  Other Names: L-leucovorin; L-leucovorin calcium; L-folinic acid, calcium salt; L-folinate, calcium salt
  Arms: L-leucovorin calcium
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the cognitive and behavioral effects of liquid leucovorin calcium on young children with autism spectrum disorder (ASD) and determine whether it improves social communication as well as the core and associated symptoms of ASD. The investigators will enroll 80 children across two sites, between the ages of 2.5 and 5 years, with confirmed ASD and known social and communication delays. Participation will last approximately 26 weeks, from screening visit to end of treatment.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a heterogeneous neurodevelopmental disorder with life-long consequences that affects young children during critical times in their development. ASD is defined by impairments in social-communication as well as the presence of restricted interests and repetitive behaviors. ASD is frequently associated with co-occurring language delays. Currently the only well-accepted treatment for core ASD symptoms is behavior therapy such as Applied Behavioral Analysis and Early Intensive Behavioral Intervention. There is no US Food and Drug Administration approved medical therapy that addresses core ASD symptoms or the pathophysiological processes that underlie ASD.

The primary aim of this study is to evaluate the effect of a liquid form of leucovorin calcium on social and communication impairments in very young children with ASD. Participants entered into the trial will have delayed language and moderate ASD symptoms. The investigators hypothesize that leucovorin calcium will significantly improve social communication as well as core and associated behavioral symptoms of ASD, and be well-tolerated with no significant adverse effects, in young children with ASD.

To assess whether the liquid form of leucovorin calcium is superior to placebo, the investigators will study 80 children across two sites, between the ages of 2.5 and 5 years, with confirmed ASD and known social and communication delays at baseline. Participants will be randomly assigned to receive active treatment or placebo for 12 weeks under double-blind conditions. At the end of 12 weeks, all participants will receive active treatment for 12 weeks. Language skills and social communication abilities will be measured at screening and after each treatment arm in order to determine if the supplement positively influences social communication. Additionally, the investigators will measure changes in neural pathways using either magnetoencephalography at Phoenix Children's Hospital or functional Near Infrared Spectroscopy at State University of New York, Downstate. While these measures will be considered exploratory, they will be important to begin to elucidate the neuronal mechanisms underlying leucovorin's impact.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Autism Spectrum Disorder (diagnosed as Autistic Disorder on the ADOS-2 or the ADI-R).
2. Between 2 years 6 months and 5 years 2 months of age at baseline
3. Folate Receptor Alpha Autoantibody Positive status
4. Language impairment (Ages and Stage Questionnaire between -1 and -3 SD for Language)
5. English included in the languages in which the child is being raised
6. Autism severity of moderate or higher (≥4) under the 7-item clinical global impression-severity scale. Moderate level of autism severity (4) is defined by the diagnosis of ASD with language impairment, so fulfilling #1 and #4 fulfills this requirement.
7. Ability to maintain all ongoing complementary, dietary, traditional, and behavioral treatments constant for the study period
8. Unchanged complementary, dietary, traditional, and behavioral treatments for two months prior to study entry
9. Has at least 4 month old expressive language ability as assessed by the MSEL Expressive Language Scale (i.e., Parent answers "yes" to " Voluntary babbling (such as 'bu, bu, bu")" Question #7 on the MSEL Expressive Language Scale.
10. Ability to attend to social stimulus and tolerate imaging procedures, as determined at the discretion of the investigator

Exclusion Criteria:

1. Known FRAA status by clinically validated test performed outside of research studies.
2. Mineral or vitamin supplementation that exceeds the Tolerable Upper Daily Intake Levels set by the Institute of Medicine (See Table 6 below)
3. Significant self-abusive or violent behavior or evidence of suicidal ideation, plan or behavior
4. Severely affected children as defined by CGI-Severity Standard Score = 7 (Extremely Ill)
5. Severe prematurity (<34 weeks gestation) as determined by medical history
6. Current uncontrolled gastroesophageal reflux
7. Current or history of liver or kidney disease as determined by medical history and safety labs
8. Genetic syndromes
9. Congenital brain malformations
10. Epilepsy
11. Any medical condition that the PI determines could jeopardize the safety of the study subject or compromise the integrity of the data
12. Significant negative reaction (i.e. fainting, vomiting, etc.) as a result of a previous blood draw.
13. Failure to thrive or Body Mass Index < 5%ile or <5%ile for weight (male <11.2kg; female <10.8kg by CDC 2000 growth charts) at the time of the study.
14. Concurrent treatment with drug that would significantly interact with l-leucovorin such as specific chemotherapy agents, antimalarial and immune suppressive agents and select antibiotics (See Table 7 below).
15. Allergy or Sensitivity to ingredients in the investigational product or placebo
16. Evaluation with the MSEL or BOSCC within 3 months of entering the study
17. Planned evaluation with the MSEL or BOSCC during the study
18. Exclusion Criteria for the MEG recording include:

    1. Ferromagnetic implants, artificial joints, fixation hardware, dental work or shrapnel (additional screening will be completed to determine MRI eligibility)
    2. Ferromagnetic products attached to the body (including hair extensions)
    3. Head circumference greater than 60 cm
    4. A weight greater than 407 lbs. (185 kg)

Ages: 30 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change in social communication symptoms | Baseline, Week 6, Week 12, Week 24
  Aberrant Behavior Checklist-2, Social Withdrawal Subscale. The ABC is a 58-item parent-reported measure with ratings in the following domains: irritability, social withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech. Each item is rated from 0 (Not a Problem) to 3 (Severe Problem). The raw score will be reported. The total raw score is the sum of the domain raw scores. A higher raw score in any of the domains indicates more severe problems in that domain; a higher total raw score indicates more severity of stereotypical autism symptoms overall.

SECONDARY OUTCOMES:
Evaluate the safety and tolerability of L-leucovorin calcium in young children with ASD | Screening, Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12, Week 16, Week 20, Week 24
  Modified Dosage Record and Treatment Emergent Symptoms: treating clinician will perform a review of medical and behavioral history at each visit to assess incidence of treatment-emergent adverse events. The treating clinician will use the scale to record presence and intensity of adverse effects. Intensity is rated on a scale of 0 (Not present) to 3 (Severe). The treating clinician will also judge the adverse effects' relatedness to treatment. Relatedness is rated on a scale of 1 (None) to 4 (Defined). The treating clinician will denote action taken. Action taken is rated on a scale of 0 (None) to 5 (Discontinue Treatment). No total score is calculated. However, higher ratings on any individual item indicate greater severity of adverse effects.
Evaluate adverse effect symptoms in young children with ASD | Screening, Week 12, Week 24
  Routine complete blood counts will be collected to determine whether treatment-emergent basic blood chemistry is altered. Presence of any changes during the course of study enrollment will be evaluated by the treating physician and determined clinically significant or not clinically significant. If determined by the treating physician, a change will be considered an adverse event.
Evaluate the biologic safety of L-leucovorin calcium in young children with ASD | Screening, Week 12, Week 24
  Routine comprehensive blood panels will be collected to determine whether treatment-emergent basic blood chemistry is altered. Presence of any changes during the course of study enrollment will be evaluated by the treating physician and determined clinically significant or not clinically significant. If determined by the treating physician, a change will be considered an adverse event.
Evaluate the safety of L-leucovorin calcium in young children with ASD on antiepileptic drugs | Screening, Week 12, Week 24
  For children using antiepileptic drugs, the level of that drug will be measured. If determined by the treating physician, a change will be considered an adverse event.
Examine the change in measures of Expressive and Receptive Language | Baseline, Week 12, Week 24
  Mullen Scales of Early Learning: a scale of cognitive abilities across core domains: visual reception, fine motor, expressive language, receptive language. Expressive language domain: 28-item scale with a raw score range of 0-50, t score range of 20-80. Receptive language domain: 33-item scale with a raw score range of 0-48, t score range of 20-80. Change in domain ability will be measured by the change in domain raw and t score. T scores are calculated from raw scores and based on age norms. A higher domain t score indicates a higher level of ability in that domain.
Evaluate the change in effects of autism symptoms on family members | Baseline, Week 6, Week 12, Week 24
  Parent Target Problems: a parent-nominated list of 2 most problematic core autism symptoms. Responses are documented in a brief narrative and detail frequency, constancy, intensity, and impact of behavior on the family. Subjective reports of frequency, constancy, intensity, and impact on family will be rated by a blinded statistician at the conclusion of the study. Higher scores indicate more severe impact on family.
Evaluate the change in stereotypical autism symptoms | Baseline, Week 6, Week 12, Week 24
  Aberrant Behavior Checklist-2: a 58-item parent-reported measure of stereotypical autism behaviors with ratings in the following domains: irritability, social withdrawal, stereotypic behavior, hyperactivity, and inappropriate speech. Each item is rated from 0 (Not a Problem) to 3 (Severe Problem). The raw score will be reported. The total raw score is the sum of the domain raw scores. A higher raw score in any of the domains indicates more severe problems in that domain; a higher total raw score indicates more severity of stereotypical autism symptoms overall.
Evaluate change in overall autism severity | Baseline, Week 6, Week 12, Week 24
  Clinical Global Impression Scale: The Clinical Global Impression Scale-Severity is a 7-point measure of overall symptom severity, ranging from 1 (Normal) to 7 (Extreme), with a raw score range of 1-7. The raw score will be reported. The Clinical Global Impression Scale-Improvement is a measure in change of symptom severity, ranging from 1 (Very Much Improved) to 7 (Very Much Worse). A Score of 4 indicates no change in symptom severity.
Evaluate change in specific autism symptom severity | Baseline, Week 6, Week 12, Week 24
  Ohio State University Clinical Impressions Scale: a clinical rating of severity and improvement of 10 autism domains: social interaction, aberrant/abnormal behavior, repetitive/ritualistic behavior, verbal communication, non-verbal communication, hyperactivity/inattention, anxiety/fears, sensory sensitivities, restricted/narrow interests, autism. Severity will be measured at baseline. Each item is rated from 1 (Normal) to 7 (Among the most severe) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment. At the following time points, improvement will be measured. Each item is rated from 1 (Very much improved) to 7 (Very much worse) with a raw score range of 10-70. The raw score will be reported. Higher scores indicate more severe impairment.
Evaluate the change in overall cognitive ability | Baseline, Week 12, Week 24
  Mullen Scales of Early Learning: a scale of cognitive abilities across core domains: visual reception, fine motor, expressive language, receptive language. Change in cognition will be measured by change in the standard Composite Scaled Score. A higher composite score indicates higher overall cognitive ability.
Evaluate the change in adaptive functioning | Baseline, Week 12, Week 24
  Vineland Adaptive Behavior Scale-II Domain Level: a scale to assess adaptive behavior in children with developmental/intellectual disabilities. This is a 135-item parent-reported measure with ratings in the following domains: communication, daily living skills, and socialization. The frequency of each item is scaled from 0 (Never) to 2 (Usually). For each domain, there are 45 items with a maximum score of 90. Change in each domain will be measured by the change in standard score. Standard scores are calculated from the raw scores and based on age norms. A higher standard score in any domain indicates a higher level of adaptive behavior in that domain. Domain standard scores will be used to get a standard composite score. Change in adaptive behavior will be measured by the change in the standard score. A higher composite score indicates higher overall adaptive behavior ability.
Evaluate the overall change in core ASD symptoms of social communication | Screening, Week 6, Week 12, Week 24
  Brief Observation of Social Communication Change: a 16-item scale that rates social interactions between children with ASD and their interactive rater. Each item is rated on a scale of 0-5, wherein 0 indicates the least severe behavior and 5 indicates the most severe behavior. A higher score is indicative of more severe social communication deficits.
Evaluate the overall change in core ASD symptoms of social communication using a blind observer | Screening, Week 6, Week 12, Week 24
  The Social Responsiveness Scale Preschool is a quantitative scale that measures severity and type of social impairments that characterize ASD. It is a standard measure in ASD clinical trials. We will use the preschool version to match the age range of our study. T-scores are calculated with a higher T-score indicating worse symptoms

OTHER OUTCOMES:
Demonstrate changes in neuronal activation and connectivity associated with treatment response using non-invasive neuroimaging methods | Baseline, Week 12, Week 24
  Using magnetoencephalography at Phoenix Children's Hospital and functional near-infrared spectroscopy and the State University of New York, the investigators will assess whether the following pathways are altered by leucovorin calcium treatment: M100 auditory evoked gamma-band power, connectivity, and coherence. Both the magnetoencephalography and functional near-infrared spectroscopy will be able to capture these same values. Treatment-emergent change in these values will indicate that a change has occurred in the neural pathway.
Evaluate the effect of L-leucovorin on cellular regulatory pathways known to be implicated in social communication | Screening, Week 12, Week 24
  Evaluate changes in the following cellular regulatory pathways known to be implicated in social communication: peripheral blood mononuclear cell, plasma, DNA, red blood cells, and oxidative stress rates. Treatment-emergent change in these biomarkers will indicate that a change has occurred at the cellular level.
Test if biomarkers (single nucleotide polymorphisms) predict clinical response to L-leucovorin | Screening, Week 12
  Saliva will be collected to determine presence of the following single nucleotide polymorphisms: MTR, MTHFR6, DHFR, GCH1, MTHFR12, RFC, FOLH, COMT. Presence or absence of these genetic polymorphisms will be analyzed to assess correlation with response to L-leucovorin treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Frye, MD, PhD, Principal Investigator — Rossignol Medical Center, Phoenix AZ
Locations (2):
- United States (2):
  - Southwestern Research & Resource Center, Phoenix, Arizona
  - State University of New York, Downstate, Brooklyn, New York

IPD SHARING:
Plan to Share IPD: No
The investigators plan to publish the results of the study in an academic journal. Results may also be shared at conferences and presentations.

REFERENCES:
- [Background] Frye RE, Rossignol DA, Scahill L, McDougle CJ, Huberman H, Quadros EV. Treatment of Folate Metabolism Abnormalities in Autism Spectrum Disorder. Semin Pediatr Neurol. 2020 Oct;35:100835. doi: 10.1016/j.spen.2020.100835. Epub 2020 Jun 25. PMID 32892962
- [Background] Frye RE, Slattery JC, Quadros EV. Folate metabolism abnormalities in autism: potential biomarkers. Biomark Med. 2017 Aug;11(8):687-699. doi: 10.2217/bmm-2017-0109. Epub 2017 Aug 3. PMID 28770615
- [Background] Frye RE, Slattery J, Delhey L, Furgerson B, Strickland T, Tippett M, Sailey A, Wynne R, Rose S, Melnyk S, Jill James S, Sequeira JM, Quadros EV. Folinic acid improves verbal communication in children with autism and language impairment: a randomized double-blind placebo-controlled trial. Mol Psychiatry. 2018 Feb;23(2):247-256. doi: 10.1038/mp.2016.168. Epub 2016 Oct 18. PMID 27752075
- [Background] Frye RE, Delhey L, Slattery J, Tippett M, Wynne R, Rose S, Kahler SG, Bennuri SC, Melnyk S, Sequeira JM, Quadros E. Blocking and Binding Folate Receptor Alpha Autoantibodies Identify Novel Autism Spectrum Disorder Subgroups. Front Neurosci. 2016 Mar 9;10:80. doi: 10.3389/fnins.2016.00080. eCollection 2016. PMID 27013943
- [Background] Frye RE, Sequeira JM, Quadros EV, James SJ, Rossignol DA. Cerebral folate receptor autoantibodies in autism spectrum disorder. Mol Psychiatry. 2013 Mar;18(3):369-81. doi: 10.1038/mp.2011.175. Epub 2012 Jan 10. PMID 22230883